CLINICAL TRIAL: NCT03800251
Title: Rate of Gastric Emptying in Term Parturients Undergoing Elective Cesarean Section
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Coombe Women and Infants University Hospital (Other)
Responsible Party: Principal Investigator, Petar Popivanov, Consultant Anaesthetist, Coombe Women and Infants University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 8-2018
Record Dates: First submitted 2019-01-06; First posted 2019-01-11 (Actual); Last update posted 2019-01-11 (Actual); Status verified 2019-01

CONDITIONS: Gastric Emptying; Pregnancy
Keywords: Gastric Emptying; Pregnancy; Elective Cesarean section; Fasting
MeSH Terms: conditions — Fasting

STUDY DESIGN:
Intervention Model Description: Patients who are fasting according to the guidelines and agree to partake in the study will, on the day of their elective LSCS, be given a 400ml carbohydrate drink at least 2hrs before their scheduled theatre time and will then have their gastric volume assessed at 15min intervals for 2hrs to determine how long it takes for the ingested fluid to leave the stomach.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fasting parturients at term (Other): Fasting parturients at term, admitted for elective cesarean section, who consent to partake in the study
  Interventions: Dietary Supplement: Nutricia PreOp - a clear, non-carbonated, lemon flavoured, carbohydrate drink that provides 0.5kcal/ml

INTERVENTIONS:
Dietary Supplement: Nutricia PreOp - a clear, non-carbonated, lemon flavoured, carbohydrate drink that provides 0.5kcal/ml — Fasting parturients at term, admitted for elective cesarean section and consent to partake in the study, will be given the intervention drink

SUMMARY:
The aim of the study is to use sequential ultrasound evaluation of the gastric volume to determine how long it takes for the stomach of a fasting pregnant woman at term, admitted for elective cesarean section, to empty after ingesting a 400ml carbohydrate drink (Nutricia preOp).

DETAILED DESCRIPTION:
Recent research suggests that attention to nutrition before operation leads to a speedier recovery through moderating the metabolic responses to surgery, improving well-being, decreasing post-operative insulin resistance and attenuation loss of lean body mass. On other hand there are fasting guidelines in place to prevent from pulmonary aspiration. The current fasting guidelines of 2hrs for clear fluids come from some small studies performed in healthy non-pregnant adults and consensus agreement.

The aim of the study is to use sequential ultrasound evaluation of the gastric volume to determine how long it takes for the stomach of a fasting pregnant woman at term, admitted for elective cesarean section, to empty after ingesting a 400ml carbohydrate drink (Nutricia preOp - a clear, non-carbonated, lemon flavoured, carbohydrate drink that provides 0.5kcal/ml).

Patients who are fasting according to the current guidelines and agree to partake in the study will, on the day of their elective LSCS, be given a 400ml carbohydrate drink at least 2hours before their scheduled theatre time. Patients will then have their gastric volume assessed at 15minutes intervals for 2 hours to determine how long it takes for the ingested fluid to leave the stomach. The results of the study will give us more information regarding gastric emptying in the investigator's patient population and may lead to reduced fasting times, increasing patient comfort and improving the patient experience.

ELIGIBILITY:
Inclusion Criteria:

* Elective LSCS
* 18yrs
* gestation >38 gestation weeks

Exclusion Criteria:

* Multiple pregnancy
* Previous upper GI surgery
* Known disorder of gastric emptying
* Hiatus Hernia
* BMI >40
* Diabetes Mellitus, Gestational Diabetes

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-06-06 (Actual); Primary Completion 2019-01 (Estimated); Study Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
Time interval required to return to the fasting grade. | 2 hours
  The stomach will be scanned and graded (Perlas grade 0-2) every 15 minutes based on the presence or absence of clear fluid in supine and right lateral decubitus position at 45 degrees elevation of the upper body, after consumption of 400 ml clear carbohydrate drink (Nutricia PreOp).

SECONDARY OUTCOMES:
Number of participants with grade 0, 1 and 2 in fasting term parturients attending for elective cesarean section | 10 minutes
  Initial "fasting" scan will be performed in all patients
Time taken for the antral cross sectional area (measured by ultrasound) to reach <9.6 cm2 (suggested cut off value for ingested volumes < 1.5ml.kg-1) after ingesting 400 ml carbohydrate drink | 2 hours
  Sequential ultrasound scans will be performed at 15 min intervals for 2 hours.
Antral cross sectional area at 2 hours | 2 hours
  Ultrasound measurement of antral cross sectional area will be performed at 2 hours after consumption of 400 ml clear carbohydrate drink (Nutricia PreOp).

CONTACTS AND LOCATIONS:
Locations (1):
- Coombe Women and Infants University Hospital, Dublin, Ireland

IPD SHARING:
Plan to Share IPD: Undecided
At the moment there is no plan whether or not to make the IPD available to other researchers.